CLINICAL TRIAL: NCT05608811
Title: The Effect of Social Skills Training on Self-efficacy, Social Phobia and Social Integration in Visually Impaired Adolescents
Brief Title: The Effect of Social Skills Training in Visually Impaired Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Esma Ozkan, Assistant Professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-187
Record Dates: First submitted 2022-10-25; First posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Visual Disorder; Young Adult; Blindness; Blindness and Low Vision; Blindness Congenital
Keywords: visually impaired; adolescent; self efficacy; social fobia; social integration
MeSH Terms: conditions — Vision Disorders; Blindness; Vision, Low

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Masking Description: Participants in the control and intervention groups were not provided with any information about which group they were in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Skills Training-intervention group (Experimental): Intervention group: Adolescents in the training group were given 8 sessions of "Social Skills Training". At the end of the training, the final evaluation was made. Initial and final assessments were made face-to-face. The training was held via Zoom.
  Interventions: Behavioral: Social Skills Training
- One Session General Social Skills-control group (Active Comparator): The control group was informed about general social skills in one session. When the training given to the intervention group was completed, the final evaluation was made. Initial and final assessments were made face-to-face.
  Interventions: Behavioral: Social Skills Training

INTERVENTIONS:
Behavioral: Social Skills Training — Intervention:
  The training is planned as 8 sessions. During this 4-week period, 2 sessions were held each week. The training, which will be held via Zoom, was carried out as a group or individual application. The first session was planned as four basic skills, the second session communication skills, the third session assertiveness skills, the fourth session conflict management skills, the fifth session social life skills, the sixth session friendship flirting skills, the seventh session health maintenance skills, and the eighth session professional/work skills.

SUMMARY:
The aim of our study is to examine the effects of eight sessions of online social skills training given to visually impaired adolescents on social skills, self-efficacy, social phobia and social integration. Forty visually impaired adolescents between the ages of 13 and 19 participated in the study. Participants were divided into control and training groups. 20 adolescents were included in the education program. All participants included in the study were evaluated using the Sociodemographic Information Form, Social Skills Assessment Scale for Children, General Self-Efficacy Scale, Child and Adolescent Social Phobia Scale, and Social Integration Questionnaire.

DETAILED DESCRIPTION:
Our study was planned to see the effect of social skills training applied to visually impaired adolescents on self-efficacy, social phobia, and social integration.

1. Inclusion Criteria:

   * Being between the ages of 13-19
   * Being visually impaired according to the health board report
   * Volunteering to participate in the study
2. Exclusion Criteria:

   * Any diagnosis or disability other than visual impairment.
   * Not understanding what you read in Turkish and what is said
   * Getting a score of ˂23 according to the Modified Mini Mental Evaluation Scale Method: In the study, a control group of 20 people and an intervention group of 20 people were formed. Individuals who met the inclusion criteria were included in the sample pool by informing them about the research. Adolescents in the training group were given 8 sessions of "Social Skills Training", while the control group was informed about general social skills in 1 session. At the end of the training, a final evaluation was made for both groups. Initial and final assessments were made face-to-face. The training was held via Zoom.

Training Plan: The training is planned in 8 sessions. During this 4-week period, 2 sessions will be held each week. The training, which will be held via Zoom, will be carried out as a group or individual application. The first session will be four basic skills, the second session will be communication skills, the third session will be assertiveness skills, the fourth session will be conflict management skills, the fifth session will be social life skills, the sixth session will be flirting friendship skills, the seventh session will be health maintenance skills. The eighth session will be about professional/work skills.

Session 1: Four Basic Skills: Listening to others, making requests, expressing positive emotions, making requests.

Session 2: Communication Skills Session 3: Assertive Skills: Refusing requests, making complaints, responding to complaints, etc.

Session 4: Conflict Management Skills Session 5: Social Life Skills Session 6: Dating and Flirting Skills Session 7: Health Maintenance Skills: Making a doctor's appointment by phone, asking about medications, asking about health-related issues, etc.

Session 8: Professional/Work Skills: Conducting job interviews, asking for feedback on job performance, etc.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 13-19
* Being visually impaired according to the health board report
* Volunteering to participate in the study

Exclusion Criteria:

* Any diagnosis other than visual impairment, presence of a disabled person
* Not understanding what you read in Turkish and what is said
* Getting a score of ˂23 according to the Modified Mini Mental Evaluation Scale

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Sociodemographic Information Form | up to one month
MESSY Children's Social Skills Assessment Scale (MESSY) | up to one month
  The scale has been developed to evaluate the social skills of children and enables the evaluation of the person regarding any sub-dimension's social skills or social status. It evaluates the sub-dimensions of Appropriate Social Skills (23 items), Inappropriate Assertiveness (21 items), Impulsivity (5 items), Self-Confidence (5 items), Jealousy/Introversion (4 items). Provides 5-point Likert type measurement. The score that can be obtained from the scale varies between 47 and 235. The validity and reliability study was carried out by Erdoğan. The scale was developed to assess children's social skills, and it enables the assessment of a person regarding any sub-dimension's social skills or social status
Child and Adolescent Social Phobia Scale | up to one month
  The scale was prepared as 35 questions in the first stage, and it was applied to 30 children with or without social phobia in the clinic, and it was checked whether the items were appropriate for the age group. Thus, some items were rearranged. Some items were removed and the number of items was reduced to 25. Provides a five-point Likert-type measurement. As the total score on the scale increases, the social phobia of individuals decreases.
General Self-Efficacy Scale | up to one month
  Sherer and his team developed together; It is a form consisting of 23 items, the validity and reliability study of which was conducted by Yıldırım and İlhan. It has 3 sub-parameters (starting-not giving up-continuation) and 17 items; It is scored according to the 5-point likert system. There is a direct ratio between the score obtained from the scale and the belief in self-efficacy, and it is possible to get a minimum of 17 and a maximum of 85 points. The reliability coefficient of the scale is 0.80 and the retest reliability coefficient is 0.69. As the total score obtained in the scale increases, the level of self-efficacy of the individuals increases.

SECONDARY OUTCOMES:
Social Integration Survey | up to one month
  The Turkish validity and reliability study was carried out by Akyürek, Salar, Bumin and Kayıhan. The validity and reliability study was conducted with the study conducted on 126 patients in the physiotherapy clinic of Ankara University Rehabilitation Hospital and Kastamonu Rehabilitation Hospital. It consists of 15 questions. As the total score on the scale increases, the social integration of the individual in the society increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Saglik Bilimleri Universitesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No